CLINICAL TRIAL: NCT07217002
Title: Reducing Antibiotic Use by Implementation of Stewardship in Primary and Urgent Care
Acronym: RAISIN
Status: Active, not recruiting | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 24-021996
Record Dates: First submitted 2025-10-09; First posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Community Acquired Pneumonia (CAP); Sinusitis; Strep Pharyngitis; Acute Otitis Media (AOM)
Keywords: Antibiotics; Antimicrobial Stewardship
MeSH Terms: conditions — Community-Acquired Pneumonia; Sinusitis; Otitis Media

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CHOP Primary Care Providers: Providers at all 31 primary care practice offices and 4 urgent care offices that include physicians and Advanced Practice Provider (APPs) including Nurse Practitioners (NPs) and Physicians Assistants (PAs).
  Interventions: Other: Online Educational Modules; Other: Prescribing Feedback Reports; Other: Clinical Decision Support; Other: Live, hybrid in-person and online educational sessions

INTERVENTIONS:
Other: Online Educational Modules — Online educational modules for clinicians that describe optimal antibiotic use and provide strategies to communicate with families about antibiotic prescribing for ARTIs. Modules are assigned through CHOP's internal learning website and assigned to every single primary care provider.
Other: Prescribing Feedback Reports — Prescribing feedback reports distributed quarterly that show clinicians how their prescribing compares to their peers and to professional guideline recommendations. Will include metrics of overall prescribing and show choice and duration for antibiotics given ear infections, Strep throat, sinus infections, and pneumonia. The goal of the feedback reports is to show clinicians how often they are prescribing antibiotics, and when they do prescribe antibiotics are they doing so with right antibiotic and for the correct duration.
Other: Clinical Decision Support — Clinical decision support built into the electronic health record to help clinicians choose the right antibiotics for the right number of days. Using information from guidelines and clinical pathways created by CHOP to help providers continue to optimize their prescribing practices.
Other: Live, hybrid in-person and online educational sessions — Live, hybrid in-person and online educational sessions that explain the project, describe best prescribing practices and allow clinicians to talk directly with project team members. Study leaders visit all 31 practices across the network.

SUMMARY:
The goal of this project is to reduce unnecessary antibiotic use for children with ARTIs (Acute Respiratory Tract Infections) by implementing "outpatient antibiotic stewardship" across the Children's Hospital of Philadelphia (CHOP) Primary and Urgent Care Network to:

1. Reduce unnecessary antibiotic prescribing for the most common infections in children.
2. Reduce unnecessary a) broad-spectrum and b) longer-course antibiotic therapy for ear infections, Strep throat, sinus infections, and pneumonia.

DETAILED DESCRIPTION:
Children often receive antibiotics for acute respiratory tract infections (ARTIs) which are caused by viruses, such as the common cold. However, antibiotics cannot treat viruses. Using antibiotics when they are not needed can cause harm - including side effects like rashes, vomiting and diarrhea - and can make it harder for the antibiotics to work when they are needed to treat infections caused by bacteria. For ARTIs caused by bacteria - like ear infections, sinus infections, strep throat or pneumonia - narrow-spectrum antibiotics are the best choice. This is because narrow-spectrum antibiotics target only the harmful bacteria, while "broad-spectrum" antibiotics target additional bacteria than can be helpful for the body. For many of these infections, it is also better to use shorter courses of antibiotics (such as five days) instead of longer courses (such as 10 days). Research studies have shown clearly that shorter courses and narrow-spectrum antibiotics cure infections just as well as longer courses and broad-spectrum antibiotics, but with fewer side effects.

Over two years, the project team will use proven strategies to ensure that children get the right antibiotics for the right amount of time. During this time, all pediatric doctors and nurse practitioners in this large, diverse network will receive:

1. Online education about proper antibiotic prescribing.
2. Regular feedback on how their antibiotic prescribing compares to peers and to professional guidelines.
3. Tools in the electronic health record to make it easy to prescribe the right antibiotics.
4. Yearly, live hybrid in-person and online educational sessions

The project team will determine how well this program works by measuring:

1. How often antibiotics are prescribed to children with ARTIs.
2. How often children with bacterial ARTIs (ear infections, sinus infections, strep throat and pneumonia) get the right antibiotic choice and right number of antibiotic days.

ELIGIBILITY:
Inclusion

* All children ages 6 months to 12 years seen at CHOP primary care network and CHOP Urgent Care with ARTI diagnoses (viral diagnoses or AOM, CAP, sinusitis, strep pharyngitis) Exclusion
* Severe immunocompromised status OR tracheostomy dependence
* Children with other bacterial infection diagnoses

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: In two years, the project team will reach all 121,000 children 6 months to 12 years of age seen at 288,000 encounters for ARTIs at the Primary Care Practices and Urgent Care locations across the CHOP primary care and urgent care network.
Sampling Method: Non-Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Antibiotic Prescribing Rates for Acute Respiratory Tract Infections (ARTIs) | From start of implementation ramp up period to end of year 2 implementation
  ARTIs as measured by overall rates of prescribing an antibiotic during clinic visits for an acute respiratory tract infection (URI) diagnosis, including both bacterial and viral URIs using the EHR. Goal is that antibiotics are prescribed at 40% or fewer ARTI visits. The optimal proportion of ARTI visits that should be associated with an antibiotic prescription is unknown. Baseline prescribing rates for antibiotics in the Network ranges from 34-61%. The target 40% rate is currently achieved by 10% of our practices with the lowest antibiotic prescribing.
Change in overall optimal antibiotic prescribing rates for all bacterial ARTI encounters | From start of implementation ramp up period to end of year 2 implementation
  Changing overall antibiotic prescribing rates as measured by a composite of 1) narrow antibiotic selection and 2) shortest effective duration as a proportion of all antibiotics prescribed for each of the target diagnoses: Acute otitis media, Group A streptococcal pharyngitis, Acute sinusitis, and Pneumonia using EHR (electronic health record) data. This metric combines both narrow-spectrum antibiotic choice and optimal durations of therapy to comprehensively evaluate optimal antibiotic prescribing. At least 90% of antibiotics prescribed for ARTI are for optimal short duration and narrow spectrum antibiotics
Broad- versus Narrow-Spectrum Antibiotic Prescribing | From start of implementation ramp up period to end of year 2 implementation
  Broad vs. Narrow-Spectrum antibiotic prescribing as measured by rates of broad-spectrum antibiotics as a proportion of all antibiotics prescribed within each of these diagnoses using the EHR (electronic health record):
  * acute otitis media
  * Group A streptococcal pharyngitis
  * acute sinusitis
  * pneumonia At least 90% of antibiotics prescribed for ARTI are for optimal narrow spectrum antibiotics.
Shortest Effective Duration Antibiotic Prescribing | From start of implementation ramp up period to end of year 2 implementation
  Shortest effective duration measured by rates of prescribing the shortest effective duration of antibiotics as a proportion of all antibiotics prescribed within each of these diagnoses:
  * acute otitis media
  * Group A streptococcal pharyngitis
  * acute sinusitis
  * pneumonia At least 90% of antibiotics prescribed for ARTI are for the shortest effective duration of antibiotics. Optimizing durations of therapy will reduce overall antibiotic days and, therefore, decrease the overall antibiotic burden for children with ARTIs.

SECONDARY OUTCOMES:
Treatment failure or modification 14 days | 14 days
  Treatment failure measured at 14 days if there is in person or telephone contact with the same ARTI diagnosis with receipt of any systemic ARTI-directed antibiotic found in the EHR. The target is for no increase in treatment failure.
Antibiotic-associated adverse events (AEs) within 7 days of completing antibiotics | From index visit to 7 days of completing antibiotics
  AEs as measured by in person or telephone contact for diarrhea, candidiasis, non-candidal rash, other or unspecified allergic reaction, other or unspecified adverse event, and vomiting using the EHR.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Same, MD, Principal Investigator — Children's Hospital of Philadelphia; Louis Bell, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided